CLINICAL TRIAL: NCT04870086
Title: A Prospective Cohort of Healthcare Workers in France
Acronym: ESPERES
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210173
Record Dates: First submitted 2021-04-08; First posted 2021-05-03 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Healthcare Workers
Keywords: Healthcare workers; Preventive measures; Attitudes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ESPERES is a national prospective e-cohort study providing a resource for collecting information on healthcare workers (HCWs) currently working in France. The overall goal of ESPERES is to develop the infrastructure necessary to create and engage a community of HCWs who may be eligible for participation in future research studies. ESPERES is set up to answer research questions, in the field of prevention for HCWs, prevention for their own health, that of their relatives, their colleagues, and users of the hospital. These research questions will be carried out in the context of specific subsequent studies. The first study that will be carried out is related to prevention against COVID-19, in particular vaccination against COVID-19 and more broadly on the COVID-19 pandemic.

DETAILED DESCRIPTION:
The study population will be made up of HCWs. For the purposes of this study, a "healthcare worker" is defined as an individual who currently works in a setting where individuals receive healthcare (i.e. individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as administrative office, housekeeping, food service, etc.). ESPERES will be offered to all the HCWs of the Assistance Publique - Hôpitaux de Paris (AP-HP) establishments and to other public or private health establishments (lucrative or not) in the Ile-De-France region and to establishments in other French regions, in order to diversify the contexts.

Each participant is self-included and collects his own data via a web interface. This cohort is open, meaning that eligible people can be included until the end of the study (no limited inclusion period). This cohort will start in 2021 and is scheduled for an initial duration of 24 months but may be extended as part of amendments.

Participants will be regularly asked to answer online questionnaires lasting at most 20 minutes. The frequency of these questionnaires will not exceed one questionnaire every 2 weeks (and will generally be more spaced out). During their follow-up in the cohort, participants may be asked, depending on their characteristics, to participate in studies nested in the cohort.

All data from ESPERES will be gathered in a health data repository. The statistical analyses planned in the research protocol and those responding to specific subsequent studies nested in ESPERES and validated by the scientific committee, will be performed by the pharmaco-epidemiology center (CEPHEPI), under the responsibility of Dr Candice ESTELLAT and Pr Florence TUBACH. The CEPHEPI is backed by the public health department of the hospital group Pitié-Salpêtrière - Charles Foix, AP-HP.

A calculation of the sample size is not justified for this study as it aims to answer several research questions in a cohort. However, a number about 15,000 participants in ESPERES are expected.

ELIGIBILITY:
Inclusion Criteria:

* Legal age
* Healthcare workers defined as individuals who currently work in a setting where individuals receive healthcare (i.e. individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as administrative office, housekeeping, food service, etc.)
* Agreeing to participate (digital consent)

Exclusion Criteria:

- No internet access

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of HCWs. For the purposes of this study, a "healthcare worker" is defined as an individual who currently works in a setting where individuals receive healthcare (i.e. individuals do not have to work directly with patients, but may have any role within a setting where individuals receive healthcare, such as administrative office, housekeeping, food service, etc.). ESPERES will be offered to all the HCWs of the Assistance Publique - Hôpitaux de Paris (AP-HP) establishments and to other public or private health establishments (lucrative or not) in the Ile-De-France region and to establishments in other French regions, in order to diversify the contexts.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Number and percent of participants who enroll in the ESPERES cohort study by age. | Up to 24 months
Number and percent of participants who enroll in the ESPERES cohort study by health establishment. | Up to 24 months
Number and percent of participants who enroll in the ESPERES cohort study by geographic region | Up to 24 months
Number and percent of participants who enroll in the ESPERES cohort study by profession | Up to 24 months
Proportion of all participants enrolled in the ESPERES cohort study who participate in an ancillary research study | Up to 24 months
Proportion of participants who continue to supple information about their health to the ESPERES cohort study at various time points after their enrollment | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence Tubach, MD, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière - Charles Foix, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ricci L, Fery C, Tubach F, Agrinier N, Gagneux-Brunon A. Health care institutions and their physicians are the greatest promoters of COVID-19 vaccine acceptance among health care workers. Vaccine. 2025 Apr 30;54:127005. doi: 10.1016/j.vaccine.2025.127005. Epub 2025 Mar 14. PMID 40088510